CLINICAL TRIAL: NCT04524455
Title: A Phase 1b Open-label Study Investigating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Administration of Blinatumomab in Combination With AMG 404 for the Treatment of Adults With Relapsed or Refractory B Cell Precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Blinatumomab in Combination With AMG 404 for the Treatment of Adults With Relapsed or Refractory B Cell Precursor ALL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190177
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Blinatumomab; AMG 404; Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab and AMG 404 (Experimental)
  Interventions: Drug: Blinatumomab; Drug: AMG 404; Drug: Dexamethasone Premedication

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab will be administered as a continuous intravenous infusion (cIV).
  Other Names: Blincyto
Drug: AMG 404 — AMG 404 will be administered as an intravenous infusion (IV).
Drug: Dexamethasone Premedication — Dexamethasone will be administered orally or intravenously prior to blinatumomab treatment, as needed.

SUMMARY:
The primary objective of this phase 1b study is to evaluate the safety and tolerability of blinatumomab and AMG 404 in combination in adults with R/R B-ALL and to estimate the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of AMG 404 when combined with continuous intravenous infusion (cIV) blinatumomab.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years at enrollment.
* Greater than or equal to 5% blasts in the bone marrow.
* Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 2.
* Negative pregnancy test in women of childbearing potential.

Exclusion Criteria

* Cancer chemotherapy (radiotherapy, chemotherapy, antibody therapy, molecular targeted therapy) within 14 days prior to study Day 1.
* Known hypersensitivity to blinatumomab or AMG 404 or to any component of the product formulation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (19):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - University of Chicago, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Royal Melbourne Hospital, Parkville, Victoria
- Ordensklinikum Linz Elisabethinen, Linz, Austria
- France (2):
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (3):
  - Klinikum und Fachbereich Medizin Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitaetsklinikum Regensburg, Regensburg
- Italy (2):
  - Azienda Ospedaliera Universitaria di Bologna Policlinico S Orsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 22 centers in Australia, Austria, France, Germany, Italy, Netherlands, Spain, United Kingdom, and the United States between 02 October 2020 to 24 January 2023.
Groups:
- Cohort 1: Blinatumomab + AMG 404 (240 mg): Blinatumomab continuous intravenous infusion (cIV) was administered at 9 μg/day on Days 1 to 7, then at 28 μg/day thereafter. Each cycle consisted of 42 days and included a 14-day blinatumomab treatment-free interval between Days 29 and 42. The treatment-free interval could be prolonged by up to 7 days if deemed necessary by the investigator. AMG 404 was administered intravenously (IV) at 240 mg, starting on Cycle 1 Day 11 (C1D11) and dosed every 4 weeks (Q4W) thereafter. Participants could receive up to 5 cycles.
- Cohort 2a: Blinatumomab + AMG 404 (480 mg): Blinatumomab cIV was administered at 9 μg/day on Days 3 to 9, then at 28 μg/day thereafter. Cycle 1 consisted of 44 days and included a 14-day blinatumomab treatment-free interval between Days 31 and 44. Each cycle thereafter consisted of 42 days and included a 14-day blinatumomab treatment-free interval between Days 29 and 42. The treatment-free interval could be prolonged by up to 7 days if deemed necessary by the investigator. AMG 404 was administered IV at 480 mg, starting on C1D1 and dosed Q4W thereafter. Participants could receive up to 5 cycles.
Period: Overall Study
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Started | 8 | 9
Participants Who Received Blinatumomab | 8 | 8
Participants Who Received AMG 404 | 8 | 8
Completed | 4 | 3
Not Completed | 4 | 6
Not completed — Death | 3 | 3
Not completed — Decision by Sponsor | 0 | 2
Not completed — Withdrawal of Consent From Study | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Cohort 1: Blinatumomab + AMG 404 (240 mg): Blinatumomab cIV was administered at 9 μg/day on Days 1 to 7, then at 28 μg/day thereafter. Each cycle consisted of 42 days and included a 14-day blinatumomab treatment-free interval between Days 29 and 42. The treatment-free interval could be prolonged by up to 7 days if deemed necessary by the investigator. AMG 404 was administered IV at 240 mg, starting on C1D11 and dosed Q4W thereafter. Participants could receive up to 5 cycles.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg) | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (18.0) | 39.3 (15.7) | 45.7 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 6 | 6 | 12
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: Investigators determined whether an adverse event (AE) qualified as a DLT per pre-specified protocol defined criteria. An AE was defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment.
Time Frame: Cohort 1: Up to 67 days; Cohort 2a: Up to 56 days
Population: DLT Analysis Set: included DLT-evaluable participants in the Safety Analysis Set. A participant was DLT-evaluable if the participant had completed DLT-evaluable period which begins with the first AMG 404 dose and includes 28 days after the second AMG 404 dose is administered or experienced a DLT any time during the DLT-evaluable period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Number analyzed (Participants) | 3 | 7
Participants | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced Treatment-Emergent AEs (TEAEs)
Description: A TEAE was defined as any AE starting on or after first dose of blinatumomab or AMG 404. The investigator used clinical judgment to assess causal relationship. A serious AE (SAE) was defined as any AE that:
  * results in death,
  * immediately life-threatening,
  * requires in-patient hospitalization or prolongation of existing hospitalization,
  * results in persistent or significant disability/incapacity,
  * is a congenital anomaly/birth defect, and/or
  * other medically important serious AE.
  AEs of interest (EOIs) for blinatumomab included capillary leak syndrome, cytokine release syndrome, decreased immunoglobulins, elevated liver enzyme, embolic and thrombotic events, immunogenicity, infections, infusion reactions without considering duration, leukoencephalopathy, progressive multifocal leukoencephalopathy, neurologic events, neutropenia and febrile neutropenia, pancreatitis, and tumor lysis syndrome. EOIs for AMG 404 included non-infectious diarrhea and hemorrhages.
Time Frame: Median (min, max) overall duration from first dose until 30 days after last dose is: 83.4 (40.2, 274.1) days
Population: Safety Analysis Set: defined as all participants who were enrolled and received at least 1 dose of blinatumomab and AMG 404.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Number analyzed (Participants) | 8 | 8
Participants
  TEAEs | 8 | 8
  Serious TEAEs | 6 | 7
  Blinatumomab-related TEAEs | 8 | 6
  AMG 404-related TEAEs | 3 | 4
  EOIs | 8 | 8

3. Secondary Outcome: Percentage of Participants Who Achieved Complete Remission (CR) or CR With Partial Hematological Recovery (CRh) (CR/CRh)
Description: Hematological remissions were defined by the following criteria:
  CR:
  * Less than 5% blasts in the bone marrow (BM)
  * No evidence of disease
  * Full recovery of peripheral blood (PB) counts:
  * Platelets > 100 000/μl
  * Absolute neutrophil count (ANC) > 1000/μl
  CR with only CRh:
  * Less than 5% blasts in the BM
  * No evidence of disease
  * Partial recovery of PB counts:
  * Platelets > 50 000/μl and
  * ANC > 500/μl
  Percentage of participants with CR/CRh were summarized along with corresponding 95% exact confidence interval (CI) using the Clopper-Pearson method.
Time Frame: Within the first 2 cycles: Up to approximately 86 days; across all cycles: Up to approximately 274 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Number analyzed (Participants) | 8 | 8
Percentage of Participants
  Within the First 2 Cycles | 37.5 [8.5 to 75.5] | 62.5 [24.5 to 91.5]
  Across All Cycles | 37.5 [8.5 to 75.5] | 62.5 [24.5 to 91.5]

4. Secondary Outcome: Percentage of Participants Who Achieved CR
Description: Hematological remissions were defined by the following criteria:
  CR:
  * Less than 5% blasts in the BM
  * No evidence of disease
  * Full recovery of PB counts:
  * Platelets > 100 000/μl
  * ANC > 1000/μl
  Percentage of participants with CR were summarized along with corresponding 95% exact CI using the Clopper-Pearson method.
Time Frame: Within the first 2 cycles: Up to approximately 86 days; across all cycles: Up to approximately 274 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Number analyzed (Participants) | 8 | 8
Percentage of Participants
  Within the First 2 Cycles | 25.0 [3.2 to 65.1] | 50.0 [15.7 to 84.3]
  Across All Cycles | 25.0 [3.2 to 65.1] | 50.0 [15.7 to 84.3]

5. Secondary Outcome: Median Duration of CR in Participants Who Achieved CR Within First 2 Cycles
Description: Duration of CR was calculated from the date CR was first achieved within the first 2 cycles until the earliest date of disease assessment indicating a relapse event or death due to any cause, whichever occurred first. Months were calculated as days from date of CR to event/censor date, divided by 30.5.
  Median time to event and 95% CI was summarized using the Kaplan-Meier (KM) method.
Time Frame: Up to approximately 274 days
Population: Safety Analysis Set: defined as all participants who were enrolled and received at least 1 dose of blinatumomab and AMG 404. Includes only participants who achieved CR within the first 2 cycles of treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Number analyzed (Participants) | 2 | 4
Months | NA [4.4 to NA] — Median and upper CI not reached. | NA [1.6 to NA] — Median and upper CI not reached.

6. Secondary Outcome: Median Duration of CR/CRh in Participants Who Achieved CR/CRh Within First 2 Cycles
Description: Duration of CR/CRh was calculated from the date CR/CRh was first achieved within the first 2 cycles until the earliest date of disease assessment indicating a relapse event or death due to any cause, whichever occurred first. Months were calculated as days from date of CR/CRh to event/censor date, divided by 30.5.
  Median time to event and 95% CI was summarized using the KM method.
Time Frame: Up to approximately 274 days
Population: Safety Analysis Set: defined as all participants who were enrolled and received at least 1 dose of blinatumomab and AMG 404. Includes only participants who achieved CR/CRh within the first 2 cycles of treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Number analyzed (Participants) | 3 | 5
Months | NA [4.4 to NA] — Median and upper CI not reached. | NA [1.6 to NA] — Median and upper CI not reached.

7. Secondary Outcome: Steady-state Concentrations (Css) of Blinatumomab
Description: Pharmacokinetic (PK) parameters were estimated using standard non-compartmental approaches and summarized by dose level as pre-specified in the protocol.
Time Frame: Cohort 1: C1D1 and D8 (predose, 2 to 24 h postdose), and D11, D18 and D29; C2D1 (predose, 2 to 24 h postdose) and D29. Cohort 2a: C1D3 and D10 (predose, 2 to 48 h postdose), and D29, D30 and D31; C2D1 (predose, 2 to 24 h postdose), D13 and D29
Population: PK Analysis Set: Defined as all participants in the Safety Analysis Set who have at least 1 PK sample collected. Includes only participants with available data at each timepoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Cohort 1; Cycle 1: Blinatumomab 9 μg/Day: Blinatumomab cIV was administered at 9 μg/day on Days 1 to 7. Cycle 1 consisted of 42 days.
- Cohort 1; Cycle 1: Blinatumomab 28 μg/Day: Blinatumomab cIV was administered at 28 μg/day on Days 8 to 28. Cycle 1 consisted of 42 days. AMG 404 was administered IV at 240 mg, starting on C1D11 and dosed Q4W thereafter.
- Cohort 1; Cycle 2: Blinatumomab 28 μg/Day: Blinatumomab cIV was administered at 28 μg/day. Cycle 2 consisted of 42 days and included a 14-day blinatumomab treatment-free interval between Days 29 and 42. The treatment-free interval could be prolonged by up to 7 days if deemed necessary by the investigator. AMG 404 was administered IV at 240 mg, starting on C1D11 and dosed Q4W thereafter.
- Cohort 2a; Cycle 1: Blinatumomab 9 μg/Day: Blinatumomab cIV was administered at 9 μg/day on Days 3 to 9. Cycle 1 consisted of 44 days. AMG 404 was administered IV at 480 mg, starting on C1D1 and dosed Q4W thereafter.
- Cohort 2a; Cycle 1: Blinatumomab 28 μg/Day: Blinatumomab cIV was administered at 28 μg/day on Days 10 to 30. Cycle 1 consisted of 44 days. AMG 404 was administered IV at 480 mg, starting on C1D1 and dosed Q4W thereafter.
- Cohort 2a; Cycle 2: Blinatumomab 28 μg/Day: Blinatumomab cIV was administered at 28 μg/day. Cycle 2 consisted of 42 days and included a 14-day blinatumomab treatment-free interval between Days 29 and 42. The treatment-free interval could be prolonged by up to 7 days if deemed necessary by the investigator. AMG 404 was administered IV at 480 mg, starting on C1D1 and dosed Q4W thereafter.
Arm/Group | Cohort 1; Cycle 1: Blinatumomab 9 μg/Day | Cohort 1; Cycle 1: Blinatumomab 28 μg/Day | Cohort 1; Cycle 2: Blinatumomab 28 μg/Day | Cohort 2a; Cycle 1: Blinatumomab 9 μg/Day | Cohort 2a; Cycle 1: Blinatumomab 28 μg/Day | Cohort 2a; Cycle 2: Blinatumomab 28 μg/Day
Number analyzed (Participants) | 7 | 8 | 3 | 8 | 7 | 5
pg/mL | 152 (70.2) | 676 (478) | 779 (210) | 210 (177) | 638 (274) | 626 (228)

8. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 404
Description: PK parameters were estimated using standard non-compartmental approaches and summarized by dose level as pre-specified in the protocol.
Time Frame: Cohort 1: C1D11 (predose, end of infusion to 48 h postdose), D18, D29, and D39 (predose and end of infusion). Cohort 2a: C1D1 (predose, end of infusion to 168 h postdose), D12 and D29 (predose and end of infusion)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/mL
Groups:
- Cohort 1: AMG 404 (240 mg): AMG 404 was administered IV at 240 mg, starting on C1D11 and dosed Q4W thereafter. Each cycle consisted of 42 days.
- Cohort 2a: AMG 404 (480 mg): AMG 404 was administered IV at 480 mg, starting on C1D1 and dosed Q4W thereafter. Cycle 1 consisted of 44 days.
Arm/Group | Cohort 1: AMG 404 (240 mg) | Cohort 2a: AMG 404 (480 mg)
Number analyzed (Participants) | 8 | 8
mg/mL | 70.2 (18.7) | 175 (53.5)

9. Secondary Outcome: Time to Cmax (Tmax) of AMG 404
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: AMG 404 (240 mg) | Cohort 2a: AMG 404 (480 mg)
Number analyzed (Participants) | 8 | 8
Hours | 2.5 [0.45 to 25] | 1.5 [0.50 to 2.8]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 28 Days Post Infusion (AUC0-28d) of AMG 404
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: day·mg/mL
Arm/Group | Cohort 1: AMG 404 (240 mg) | Cohort 2a: AMG 404 (480 mg)
Number analyzed (Participants) | 7 | 8
day·mg/mL | 750 (269) | 1920 (660)

11. Secondary Outcome: Number of Participants With Incidences of Anti-Blinatumomab Antibodies
Description: Only samples testing positive for anti-blinatumomab binding antibodies were to be tested for neutralizing antibodies (NAbs) as pre-specified in the protocol.
Time Frame: Up to approximately 274 days
Population: Safety Analysis Set: defined as all participants who were enrolled and received at least 1 dose of blinatumomab and AMG 404. Includes only participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Number analyzed (Participants) | 8 | 8
Participants
  Binding Antibody Positive at Anytime | 0 | 0
  NAb Positive at Anytime: number analyzed (Participants) | 0 | 0
  NAb Positive at Anytime | 0 | 0

12. Secondary Outcome: Number of Participants With Incidences of Anti-AMG 404 Antibodies
Description: Only samples testing positive for anti-AMG 404 binding antibodies were to be tested for NAbs as pre-specified in the protocol.
Time Frame: Up to approximately 274 days
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
Number analyzed (Participants) | 8 | 8
Participants
  Binding Antibody Positive at Anytime | 0 | 0
  NAb Positive at Anytime: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs: median (min, max) overall duration from first dose until 30 days after last dose is: 83.4 (40.2, 274.1) days. All-cause mortality: median (min, max) overall duration from enrolment until end of study is 152 (7, 360) days.
Description: All-cause mortality was collected for all participants enrolled/randomized in the study. Serious AEs and other AEs were collected for all participants who received at least one dose of study drug.
Arm/Group | Cohort 1: Blinatumomab + AMG 404 (240 mg) | Cohort 2a: Blinatumomab + AMG 404 (480 mg)
All-Cause Mortality (participants affected / at risk) | 3/8 | 3/8
Serious Adverse Events (participants affected / at risk) | 6/8 | 7/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Blinatumomab + AMG 404 (240 mg) (N=8) | Cohort 2a: Blinatumomab + AMG 404 (480 mg) (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Condition aggravated (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Blinatumomab + AMG 404 (240 mg) (N=8) | Cohort 2a: Blinatumomab + AMG 404 (480 mg) (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 2
Deafness (Ear and labyrinth disorders) | 2 | 0
Dry eye (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 4 | 0
Asthenia (General disorders) | 1 | 2
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Generalised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 3 | 0
Pyrexia (General disorders) | 7 | 4
Swelling (General disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 3 | 3
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Puncture site cellulitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood lactate dehydrogenase decreased (Investigations) | 1 | 0
Blood lactic acid increased (Investigations) | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Immunoglobulins decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Vascular purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT04524455/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT04524455/SAP_001.pdf